CLINICAL TRIAL: NCT05544838
Title: Simulation Based Comparison Of Standard Versus Rotational Laryngeal Mask Airway Insertion Technique In Novice Anesthesiologists. A Randomised Control Crossover Trial
Brief Title: Simulated Comparison of Standard Versus Rotational Laryngeal Mask Airway Insertion in Novice Anaesthesiologists.
Acronym: LMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dileep Kumar, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2022-6256-22361
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Training Group, Sensitivity
Keywords: LMA; Technique; Standard; Rotational; Simulation
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Each novice resident will place ten times LMA insertion with each insertion technique in randomised cross over manner by dividing the residents in two groups (5 residents in each group), by draw method. The one group will place LMA with standard insertion technique and other group will place by rotational LMA insertion technique, then after, the groups will switch over with concerned insertion techniques
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LMA with standard insertion technique (No Intervention): Standard LMA insertion technique; LMA held like a pen and index finger placed at the junction of LMA tube and cuff. Index finger used to press LMA against hard palate and posterior pharyngeal wall until definite resistance felt at the base of hypopharynx. LMA then held with non- dominant hand and index finger removed.
- Rotational LMA insertion technique (Experimental): Rotational LMA insertion; LMA inserted like guedel airway insertion: LMA proximally grasped close to anaesthesia circuit attachment. Insertion was conducted with LMA cuff facing towards nose, hard palate and then advanced into the base of hypopharynx until resistance was felt. At this point, LMA rotated at 180 degree anti-clockwise and LMA tube black line positioned and confirmed on the nasal side.
  Interventions: Device: LMA insertion with standard technique

INTERVENTIONS:
Device: LMA insertion with standard technique — Standard LMA insertion technique; LMA held like a pen and index finger placed at the junction of LMA tube and cuff. Index finger used to press LMA against hard palate and posterior pharyngeal wall until definite resistance felt at the base of hypopharynx. LMA then held with non- dominant hand and index finger removed.
  Rotational LMA insertion; LMA inserted like guedel airway insertion: LMA proximally grasped close to anaesthesia circuit attachment. Insertion was conducted with LMA cuff facing towards nose, hard palate and then advanced into the base of hypopharynx until resistance was felt. At this point, LMA rotated at 180 degree anti-clockwise and LMA tube black line positioned and confirmed on the nasal side.
  Other Names: Rotational LMA insertion technique
  Arms: Rotational LMA insertion technique

SUMMARY:
The primary objective of study was to compare insertion ease by standard and rotational LMA insertion technique on basis of LMA insertion attempts and insertion time duration. The secondary objective of study was to analyse impact of prior information for airway device, insertion techniques, general or specific work experience in airway management with ease of both insertion techniques. And, tertiary objective of study was to analyse the trainee's preference insertion technique on basis of learning method and practical adaptability.

Hypothesis:

The rotational LMA insertion technique is easy to understand and practice than the standard LMA insertion technique at the beginning of airway management training among the novice anesthesiologists.

Hypothesis:

The rotational LMA insertion technique is easy to understand and practice than the standard LMA insertion technique at the beginning of airway management training among the novice anesthesiologists.

DETAILED DESCRIPTION:
* LMA insertion attempts are the number of LMA insertion attempts with each study's insertion technique. The 10 insertion attempts will be performed with each insertion technique by trainees.
* LMA insertion time duration is the time taken to complete LMA insertion; from the holding of device till the confirmation of chest movement (artificial lungs inflation in manikin).
* The correlation of previous information for airway device, insertion techniques, general or specific work experience in airway management with the ease of both study's insertion techniques will be asked by participant's through the questionnaire at the start of study.
* The trainees will be asked at the end of study for preferred insertion method at novice level on the basis of learning method and practical conduct (user friendly)

ELIGIBILITY:
Inclusion Criteria:

* First year anaesthesia trainee
* Using adult mannequin

Exclusion Criteria:

* Paediatric mannequin
* Participant's refusal

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2021-10-02 (Actual); Study Completion 2021-10-02 (Actual)

PRIMARY OUTCOMES:
The ease of LMA insertion was measured on the basis of number of LMA insertion attempts. | 5 minute
  Ease of LMA insertion in mannequin mouth was measured by performing the 10 times insertion of LMA with both study techniques in mannequin mouth by trainees.
The ease of LMA insertion was measured on the basis of final LMA insertion time taken duration. | 5 minutes
  The total time duration of final LMA insertion confirmation in mannequin mouth was recorded. The time duration counting was started from LMA holding in operator's hand to the confirmed successful insertion in mannequin mouth.

SECONDARY OUTCOMES:
The trainee's baseline knowledge was assessed for the type of supraglottic airway devices and LMA insertion techniques. | 1 minute
  The questionnaire based trainee's asked for the prior information of the LMA and other supraglottic airway devices.
The trainee's baseline knowledge was assessed for the type LMA insertion techniques. | 1 minute
  The trainee's baseline knowledge was assessed for the type LMA insertion techniques.
The trainee's baseline knowledge was assessed for the general or specific work experience in airway management using the LMA. | 1 minute
  The questionnaire based trainee's asked for previous experience in using the LMA device.
The trainee's baseline knowledge was assessed for the studied Rotational LMA insertion technique. | 2 minutes
  The questionnaire based trainee's asked for the previous experience for rotational LMA insertion technique.

OTHER OUTCOMES:
The trainee's asked for the choice of LMA insertion technique at the start of learning airway management using the LMA device at his level. | 2 minutes
  The questionnaire based trainee's asked for the choice of type of LMA insertion technique such as standard or rotational LMA insertion at start of learning the airway management at his level of training year.
The trainee's asked for the easy learning of LMA insertion technique at his level of training. | 2 minutes
  The questionnaire based trainee's asked for his experience of easy learning of type of LMA insertion technique such as standard or rotational LMA insertion at his level of training year.
The trainee's asked for the preference of LMA insertion technique in his practice at his level of training. | 1 minute
  The questionnaire based trainee's asked for his preference to practice most of the time for the type of LMA insertion technique like standard or rotational LMA insertion at his level of training year.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The plan is to publish the study and consent has been taken from participants.
Supporting Information: SAP, CSR
Time Frame: Data is available
Access Criteria: Through publication only
URL: http://www.aku.edu

REFERENCES:
- [Background] Kumar D, Khan M, Ishaq M. Rotational vs. standard smooth laryngeal mask airway insertion in adults. J Coll Physicians Surg Pak. 2012 May;22(5):275-9. PMID 22538029
- [Background] Komasawa N, Berg BW. Simulation-based Airway Management Training for Anesthesiologists - A Brief Review of its Essential Role in Skills Training for Clinical Competency. J Educ Perioper Med. 2017 Oct 1;19(4):E612. eCollection 2017 Oct-Dec. PMID 29766036
- [Background] Kennedy CC, Cannon EK, Warner DO, Cook DA. Advanced airway management simulation training in medical education: a systematic review and meta-analysis. Crit Care Med. 2014 Jan;42(1):169-78. doi: 10.1097/CCM.0b013e31829a721f. PMID 24220691
- [Background] Lee DW, Kang MJ, Kim YH, Lee JH, Cho KW, Kim YW, Cho JH, Kim YS, Hong CK, Hwang SY. Performance of intubation with 4 different airway devices by unskilled rescuers: manikin study. Am J Emerg Med. 2015 May;33(5):691-6. doi: 10.1016/j.ajem.2015.03.006. Epub 2015 Mar 12. PMID 25800412
- [Result] Liti A, Giusti GD, Gili A, Giontella M, Dell'Omo S, Camerlingo V, Fronteddu A, Galazzi A, Bambi S. Insertion of four different types of supraglottic airway devices by emergency nurses. A mannequin-based simulation study. Acta Biomed. 2020 Nov 30;91(12-S):e2020016. doi: 10.23750/abm.v91i12-S.10832. PMID 33263351
- [Derived] D K, C K. Simulation-Based Comparison of Standard Versus Rotational Laryngeal Mask Airway Insertion Techniques in Novice Anesthesiologists: A Randomized Controlled Crossover Trial. Anesthesiol Res Pract. 2025 Dec 31;2025:7850095. doi: 10.1155/anrp/7850095. eCollection 2025. PMID 41479467